CLINICAL TRIAL: NCT07391007
Title: A Multidimensional Early-Recurrence Risk Stratification System and Personalized Treatment for Colorectal Cancer Liver Metastases: A Prospective Clinical Study
Brief Title: Integrated Clinical-molecular Risk Stratification to Early Recurrence in Colorectal Liver Metastases
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yibin Wu, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: 2025-Exp196-KY
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Liver Metastases
MeSH Terms: interventions — Base Sequence; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor sample tissues from liver metastatic lesions and poseoperative blood samples at month 1 (before adjuvant chemotherapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FUSCC Prospective Cohort: FUSCC Prospective Cohort
  Interventions: Other: gene sequencing; Other: observational study

INTERVENTIONS:
Other: gene sequencing — All patients will be performed gene sequencing in this study
Other: observational study — Observational Study

SUMMARY:
The goal of this observational study is to develop an integrated clinical-molecular risk stratification to identifypatients who are at high risk of recurrence and who would benefit from adjuvant chemotherapy in patients with recectable colorectal liver metastases. The main question it aims to answer is: can the integration of multi-dimensional data-including ctDNA, driver gene profiles, and clinical factors-accurately identify postoperative patients at high risk of recurrence and guide personalized adjuvant therapy strategies?

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, inclusive (male or female).
2. Pathologically and radiologically confirmed colorectal cancer with liver metastases.
3. Must have undergone complete (R0) surgical resection of both the primary colorectal tumor and all liver metastases.
4. Have adequate organ function and no contraindications to potential adjuvant therapies (surgery, chemotherapy, radiotherapy, immunotherapy).
5. Willing and able to comply with the study protocol and follow-up visits.
6. Availability of sufficient liver metastasis tumor tissue for gene sequencing.
7. Provision of a blood sample for circulating tumor DNA (ctDNA) detection within one month after surgery but before starting any adjuvant therapy.

Exclusion Criteria:

1. Pregnancy or breast-feeding women
2. History of other malignancies within 5 years (except cured skin cancer and cervicalcancer in situ)
3. History of uncontrolled epilepsy, central nervous system disease, or psychiatricdisorders
4. Clinically serious heart disease, such as symptomatic coronary artery disease, NewYork Heart Association (NYHA) class II or worse congestive heart failure or severearrhythmia requiring pharmacologic intervention, or history of myocardial infarctionwithin the last 12 months
5. Baseline blood and biochemical indicator do not meet the following criteria:neutrophils >=1.5×10^9/L, Hb >=90g/L, PLT >=100×10^9/L, ALT/AST<=2.5 ULN, Cr <= 1ULN
6. Allergic to any component of the therapy
7. Severe uncontrolled recurrent infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with resectable colorectal liver metastases
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Model Performance | 2-years
  We used the area under the ROC curve (AUC) and calibration curves to evaluate the predictive performance of the model.
2-year recurrence free survival | From enrollment to the end of recurrence at 2 years

SECONDARY OUTCOMES:
3-years overall survival | From enrollment to the end of death at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The ownership and usage rights of the data from this study are subject to agreements with the participating institutions, funding organizations, and sample providers. These agreements stipulate that the data may only be used for the specific purposes of this project and, therefore, cannot be publicly shared.

REFERENCES:
- [Result] Faulkner LG, Howells LM, Pepper C, Shaw JA, Thomas AL. The utility of ctDNA in detecting minimal residual disease following curative surgery in colorectal cancer: a systematic review and meta-analysis. Br J Cancer. 2023 Jan;128(2):297-309. doi: 10.1038/s41416-022-02017-9. Epub 2022 Nov 8. PMID 36347967
- [Result] Wan JCM, Massie C, Garcia-Corbacho J, Mouliere F, Brenton JD, Caldas C, Pacey S, Baird R, Rosenfeld N. Liquid biopsies come of age: towards implementation of circulating tumour DNA. Nat Rev Cancer. 2017 Apr;17(4):223-238. doi: 10.1038/nrc.2017.7. Epub 2017 Feb 24. PMID 28233803
- [Result] Imai K, Allard MA, Benitez CC, Vibert E, Sa Cunha A, Cherqui D, Castaing D, Bismuth H, Baba H, Adam R. Early Recurrence After Hepatectomy for Colorectal Liver Metastases: What Optimal Definition and What Predictive Factors? Oncologist. 2016 Jul;21(7):887-94. doi: 10.1634/theoncologist.2015-0468. Epub 2016 Apr 28. PMID 27125753
- [Result] Moretto R, Germani MM, Borelli B, Conca V, Rossini D, Boraschi P, Donati F, Urbani L, Lonardi S, Bergamo F, Cerma K, Ramondo G, D'Amico FE, Salvatore L, Valente G, Barbaro B, Giuliante F, Di Maio M, Masi G, Cremolini C. Predicting early recurrence after resection of initially unresectable colorectal liver metastases: the role of baseline and pre-surgery clinical, radiological and molecular factors in a real-life multicentre experience. ESMO Open. 2024 Apr;9(4):102991. doi: 10.1016/j.esmoop.2024.102991. Epub 2024 Apr 16. PMID 38631269
- [Result] Canellas-Socias A, Sancho E, Batlle E. Mechanisms of metastatic colorectal cancer. Nat Rev Gastroenterol Hepatol. 2024 Sep;21(9):609-625. doi: 10.1038/s41575-024-00934-z. Epub 2024 May 28. PMID 38806657